CLINICAL TRIAL: NCT01136941
Title: Phase I Trial of Zileuton CR in Children and Adults With Sickle Cell Disease
Brief Title: Trial of Zileuton CR in Children and Adults With Sickle Cell Disease
Acronym: Zileuton
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-1622
Record Dates: First submitted 2010-05-13; First posted 2010-06-04 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — zileuton

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Research participants will be administered Zileuton according to the dose escalation/de-escalation schema provided in the protocol.
  Interventions: Drug: Zileuton

INTERVENTIONS:
Drug: Zileuton — Zileuton is available as a 600 mg tablet. Dosing begins at 2.4gm/day and will be increased to 3.0gm/day. Tablets will be taken twice daily for the 6 week duration of the study.

SUMMARY:
The purpose of this research study is to test the safety of Zileuton and see what effects (good and bad) it has on you, other children and adults with Sickle Cell Disease (SCD). The investigators also want to see how Zileuton is handled by your body at different doses.

Zileuton is a drug that is approved by the Food and Drug Administration (FDA) for the treatment of asthma for people age 12 and older. The FDA has not approved Zileuton for the treatment of SCD, so it is being studied as an investigational drug for SCD through an application to the FDA. In asthma patients, Zileuton helps by reducing inflammation. This study will see if Zileuton helps to reduce inflammation associated with SCD.

DETAILED DESCRIPTION:
Inflammation is now recognized as central to the pathophysiology of sickle cell disease (SCD), and is manifest as leukocytosis, elevated levels of inflammatory cytokines, and activation of monocytes, polymorphonuclear leukocytes (PMN) and endothelial cells. It is present at steady state and is strongly associated with acute events, acute chest and early mortality. Inflammation contributes to endothelial cell dysfunction, potentiates vaso-occlusion, and may also give rise to the airway hyper-reactivity (AHR) that often accompanies SCD. A spectrum of lung disease is seen in this patient population, from AHR and obstructive lung disease in children, to restrictive lung disease and pulmonary vascular remodeling in adults.

Evidence from our laboratory suggests that a specific angiogenic cytokine, Placenta Growth Factor that is produced by hyperplastic erythroid marrow cells and elevated in SCD, contributes to activation of monocytes and endothelial cells by inducing a key leukotriene (LT) synthetic enzyme, 5-Lipoxygenase (5LO). 5LO increases production of LT. LT are among the most potent inflammatory mediators known. LT-B4 is a very potent chemoattractant and activator of PMN and enhances endothelial cell activation, and cysteinyl LT produce airway smooth muscle constriction and inflammation in lung. Elevated LT-B4 and cysteinyl LT, and a high incidence of AHR are observed in patients with SCD. Zileuton (ZL) is a specific inhibitor of 5LO that decreases LT production, and is FDA-approved for treatment of asthma for individuals 12 years of age or older. In the context of SCD, ZL reduced adhesion of PMN and sickle RBC to rat pulmonary vasculature. In vitro data shows that ZL also increased fetal hemoglobin (HbF) production from erythroid cells in vitro, and could have additive/synergistic effects with hydroxyurea (HU). Thus, ZL may be beneficial in SCD by reducing inflammation, mitigating AHR, and increasing HbF.

We hypothesize that inhibition of 5LO activity with ZL will be safe, feasible; will significantly reduce leukotrienes and biomarkers of inflammation, will decrease AHR; and will induce HbF in patients with SCD.

We will test this hypothesis in a Phase I study of ZL in SCD. First, we will establish a safe dose of ZL and its pharmacokinetics in patients with SCD. The secondary objectives will be to determine its pharmacodynamic effects on biological endpoints and compliance to twice daily ZL administration.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SCD (HbSS,HbSC,HBS Beta thalassemia, or HBS 0 thalassemia)
* Absence of an acute sickle event or ACS in the last 4 wks
* Not on hydroxyurea
* Ability to swallow pills
* Ability to comply with pulmonary function testing

Exclusion Criteria:

* History of active hepatitis
* HIV positivity
* Pregnant or nursing
* Unable to comply with contraceptive measures
* On an investigational drug within 4 weeks
* On hydroxyurea, leukotriene antagonists (e.g., Singulair) or steroids, theophylline, coumadin, terfenadine or beta-2 blockers that affect the airway: carteolol, carvedilol, labetalol, nadolol, penbutolol, pindolol, sotalol and timolol, or on propranolol for the last four weeks
* On chronic transfusion therapy
* A serious, concurrent illness that would limit ability to complete or comply with the study requirements
* Males who drink alcoholic beverages >5-6 drinks/day or females who drink alcoholic beverages >3-4 drinks/day

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Adverse Event Grading as a Measure of Safety and Tolerability | Outcome measures will be assessed at all study visits. Visits occur at week 1, Week 2, Week 4 and Week 6. Follow-up assessments will take place at Weeks 8 and 10.
  The drug will be considered safe and tolerable if there is no grade-4 toxicity and no irreversible grade-3 toxicity upon de-escalation or discontinuation. The dose for the Part 2 portion of the trial will be the dose at which there was no DLT in 5 out of 6 at highest dose level below the maximally administered dose.
Characterization of the Distribution of Zileuton Pharmacokinetic Parameter Estimates and Drug Exposure | Outcome measures will be assessed at study visits occurring at Visit 1, week 1, Week 2, Week 3 and Week 5.
  We do not anticipate a difference in PK from normal controls. PK analysis will be performed to verify steady state levels of ZL and LT are similar to normal controls.

CONTACTS AND LOCATIONS:
Overall Officials: Punam Malik, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States